CLINICAL TRIAL: NCT06439927
Title: Nasal Septal Perforation Closure Using a 3-dimensional Fabricated Polycaprolactone Nasal Mesh
Brief Title: New Method to Close Nasal Septal Perforation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Hossam Sebaey, Assistant lecturer of otorhinolaryngology, Helwan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: self sponsored
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Nasal Perforated Septum
Keywords: nasal septal perforation
MeSH Terms: conditions — Nasal Septal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polycaprolactone nasal mesh (Experimental)
  Interventions: Device: Polycaprolactone nasal mesh

INTERVENTIONS:
Device: Polycaprolactone nasal mesh — a 3-dimensional fabricated Polycaprolactone nasal mesh

SUMMARY:
The goal of this clinical trial is to investigate if a 3-dimensional fabricated nasal mesh works to close nasal septal perforations. Under general anesthesia, during nasal septal perforation repair surgery, the investigator will place the mesh between the elevated mucoperichondrial flaps opposite the site of the perforation and confirm its original position at both sides under nasal endoscope. Endoscopic examination for septal mucosa status will be done monthly for a three months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing nasal septal perforation repair surgery.

Exclusion Criteria:

* Patients with known allergy to polycaprolactone.
* Pregnancy or lactation.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Post-operative healing of septal perforation | for a three months follow up period
  Endoscopic evaluation of nasal septal mucosa status will be classified as complete bilateral healing, complete unilateral healing, no healing, and perforation.

SECONDARY OUTCOMES:
Postoperative complications | for a three months follow up period
  The following complications will be evaluated on a present/absent basis:hematoma-infection-allergy

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Sebaey, master degree, Principal Investigator — Helwan University
Locations (1):
- Faculty of Medicine, Helwan University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No